CLINICAL TRIAL: NCT03927781
Title: Perioperative Pregabalin as Part of a Multimodal Treatment Plan for Pain After Ureteroscopy With Stent Placement: a Pilot
Brief Title: Perioperative Pregabalin in Ureteroscopy: a Pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Katie Murray, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013680
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Nephrolithiasis; Urolithiasis; Perioperative/Postoperative Complications; Pain, Postoperative; Pain, Acute; Anesthesia; Urologic Diseases; Anesthesia Morbidity
Keywords: Pregabalin; Perioperative medicine; Opioid sparing; Urolithiasis; Ureteroscopy
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis; Postoperative Complications; Pain, Postoperative; Acute Pain; Urologic Diseases | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: All participants will receive 300mg PO pregabalin one hour before procedure start
Masking Description: There will be no blinding for this pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pregabalin 300mg (Experimental): 300mg pregabalin, PO, once, 1 hr before surgery
  Interventions: Drug: Pregabalin 300mg

INTERVENTIONS:
Drug: Pregabalin 300mg — One 300mg capsule will be administered PO 1 hour before surgery
  Other Names: Lyrica; Gabapentinoid

SUMMARY:
The investigators propose a pilot clinical trial on the use of perioperative pregabalin in order to decrease ureteral stent related symptoms and decrease opioid usage after ureteroscopy with stent placement. Patients undergoing ureteroscopy with stent placement will receive a single dose of 300 mg pregabalin PO in the preoperative area. This work will assess safety and feasibility of studying this regimen at our institution, with the aim of performing a randomized, placebo-controlled, double-blinded study in the future.

ELIGIBILITY:
Subject Population Undergoing elective ureteroscopy with stent placement by Dr. Murray at University of Missouri Hospital and affiliated facilities

Subject Inclusion

Age >= 18 years

Subject Exclusion

* Renal insufficiency (eGFR < 30 mL/minute/1.73 m2)
* Chronic indwelling ureteral stent
* Chronic opioid use
* History of opioid abuse
* Chronic gabapentinoid use
* Plan for inpatient hospitalization
* Pregnancy
* Inability of the patient to consent for themselves in English
* Allergy to gabapentinoid
* Liver failure or hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2020-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Murray, DO, Principal Investigator — Assistant Professor
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregabalin 300mg
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 40.2 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Events Related to Study Drug
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
Participants | 6

2. Primary Outcome: Number of Participants Who Were Administered the Study Drug Correctly
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
Participants | 10

3. Primary Outcome: Respondent Reported Usability of Instruments
Description: Number of patients able to complete 30 day post op questionnaire
Time Frame: 30 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
Participants | 5

4. Secondary Outcome: Early Post-op Stent Related Symptoms
Description: Ureteral Stent Related Symptom Questionnaire (USSQ) score, sum of urinary index score, pain index score, and general health index score. Minimum is 24. Maximum is 162. Higher scores indicate a worse outcome.
Time Frame: Post-op day 3
Population: Those who completed the questionnaire
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 5
score on a scale | 88 [61 to 130]

5. Secondary Outcome: Early Post-op Opioid Needs
Description: Number of patients with a verified prescription for narcotic medication within the first 30 post-operative days.
Time Frame: First 30 post-operative days
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
Participants | 1

6. Secondary Outcome: Opioid Use
Description: Number of patients stating that they had used opioids on any survey.
Time Frame: Up to 1 year post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
Participants | 1

7. Secondary Outcome: Amount of Opioid Use
Description: Total amount of opioid used for any indication at several time points, in oral morphine equivalents. This is the sum for all patients.
Time Frame: Up to 1 year post-op
Measure: Number; unit: oral morphine equivalents
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
oral morphine equivalents | 90

8. Secondary Outcome: Unplanned Healthcare Contacts
Description: Number of unplanned contacts between the patient and the healthcare system. This is the total for all patients.
Time Frame: First 30 post-operative days
Measure: Number; unit: visits
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 10
visits | 2

9. Secondary Outcome: Patient Satisfaction
Description: Score on standardized evaluation of patient satisfaction at 7-days post-op. This was on a scale from 1) very dissatisfied to 5) very satisfied. Higher scores are better.
Time Frame: First 30 post-operative days
Population: Respondents to the survey
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Pregabalin 300mg
Number analyzed (Participants) | 6
score on a scale | 3.5 [1 to 5]

ADVERSE EVENTS:
Time Frame: Events were systematically characterized on the day of surgery. Adverse events were otherwise by report up to 30 days after the patient's procedure.
Arm/Group | Pregabalin 300mg
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 300mg (N=10)
Pain (Nervous system disorders) | 3
Increased appetite (Gastrointestinal disorders) | 1
Back pain (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 6
Fatigue (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Blurred vision (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT03927781/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03927781/SAP_001.pdf